CLINICAL TRIAL: NCT05653063
Title: ARCHERY - Artificial Intelligence Based Radiotherapy Treatment Planning for Cervical, Head and Neck and Prostate Cancer
Status: Recruiting | Type: Observational
Sponsor: University College, London (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Rising Tide Foundation (Other); Medical Research Council (Other Government); Tata Memorial Hospital (Other Government); Tata Memorial Centre (Other); University of Stellenbosch (Other); King Hussein Cancer Center (Other); University of Malaya (Other); University Ghent (Other); M.D. Anderson Cancer Center (Other); Mount Vernon Cancer Centre at Mount Vernon Hospital (Other); University of Cape Town (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: ARCHERY; 1U01CA269143-01 (NIH); 10678756 (Other: ISRCTN)
Record Dates: First submitted 2022-11-03; First posted 2022-12-16 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Cancer of Prostate; Cancer Head Neck; Cancer Cervix
MeSH Terms: conditions — Prostatic Neoplasms; Head and Neck Neoplasms; Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: A web-based artificial intelligence (AI) auto-planning tool — The CT scan taken at the time of treatment planning is uploaded to a web server called the Radiotherapy planning assistant which automates the contouring of target organs and areas of high-risk disease as well as defining the size, shape and number of radiotherapy beams to treat the cancer. The final plan is downloaded to the local treatment planning system where the doses are recalculated and clinical peer review is undertaken before the plan can be used clinically.
  In this study patients will not be treated with the AI tool but the manual plan created by the local teams.

SUMMARY:
The aim of this study is to look at whether an Artificial Intelligence (AI) based computer program can automate two components of the radiotherapy treatment pathway to a sufficient quality standard to enable its routine clinical use. The two components include the delineation (outlining) of anatomical areas that are at risk of tumour spread and at risk of radiation damage, and the definition of the position, size and shape of the radiation beams.

The AI-based computer programs have been developed to perform tasks that would normally require direct human involvement by oncologists and medical physicists. Proposed advantages include improved treatment accuracy, as well as a reduction in the time (from weeks to minutes) and human resources needed to deliver radiotherapy, which this study will test.

ELIGIBILITY:
Inclusion Criteria:

1. Consecutive patients with histologically confirmed head and neck cancers of the oropharynx, larynx, hypopharynx and nasopharynx (Stage I-III) that have given consent for radical radiotherapy.
2. Consecutive histologically confirmed primary cervical cancer patients (Stage IB-IIIB including pelvic node positive) that have given consent for radical radiotherapy.
3. Consecutive histologically confirmed primary prostate cancer patients (T1-4N0M0) that have given consent for radical radiotherapy.
4. Mental capacity to understand and consent to participate in the study.
5. Patients aged ≥18years.

Exclusion Criteria:

1. Patients requiring radiotherapy after curative surgery or surgery that is intended to remove as much of the tumour as possible.
2. Patients receiving palliative radiotherapy
3. Patients aged < 18years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients eligible for radiotherapy for head and neck, cervical or prostate cancer.
Sampling Method: Non-Probability Sample
Enrollment: 990 (Estimated)
Dates: Start 2023-12-07 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of radiotherapy treatment plans that have contours and dosimetry that meet pre-defined criteria for clinical acceptability | Prior to first treatment

SECONDARY OUTCOMES:
comparison of time and human resource requirements between producing automated radiotherapy treatment plans using artificial intelligence and producing treatment plans using the standard manual pathway | radiotherapy plan preparation process pre treatment
Comparison of radiotherapy treatment costs using the artificial intelligence automated pathway and standard manual planning pathway | radiotherapy treatment plan preparation process and treatment interval

CONTACTS AND LOCATIONS:
Locations (6):
- India (2):
  - Tata Medical Centre, Kolkata
  - Tata Memorial Hospital, Mumbai
- King Hussein Cancer Center, Amman, Jordan
- University of Malaya Medical Center, Kuala Lumpur, Malaysia
- South Africa (2):
  - Groote Schuur Hospital, Cape Town
  - Tygerberg Hospital, Stellenbosch